CLINICAL TRIAL: NCT00000583
Title: Hepatitis B Vaccine Clinical Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: 303; P01HL009011-18A1 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2012-04

CONDITIONS: Hepatitis B; Hepatitis, Viral, Human; Liver Diseases
MeSH Terms: conditions — Hepatitis B; Hepatitis, Viral, Human; Liver Diseases | interventions — Hepatitis B Vaccines

INTERVENTIONS:
Biological: hepatitis B vaccines

SUMMARY:
To determine the efficacy of a hepatitis vaccine in preventing hepatitis B.

DETAILED DESCRIPTION:
BACKGROUND:

Although most carriers of HBsAg are asymptomatic, a substantial proportion eventually develop chronic active hepatitis and cirrhosis. There is also overwhelming evidence that the hepatitis B virus is the single most important causative factor of hepatocellular carcinoma. Thus, mass immunization programs against HBV infection may ultimately affect not only the incidence of acute hepatitis B and the pool of chronic carriers but may also reduce the morbidity and mortality from chronic active hepatitis, cirrhosis, and hepatocellular carcinoma.

Krugman and his co-workers laid the groundwork for active immunization against hepatitis B in 1970 to 1973. They discovered that a 1:10 dilution of hepatitis B infective serum lost its infectivity when boiled for one minute but retained its antigenicity and prevented hepatitis B in 70 percent of vaccinated subjects. Hilleman and his colleagues at the Merck Institute of Therapeutic Research developed a more sophisticated vaccine consisting of highly purified, formalin-inactivated HBsAg particles derived from the plasma of chronic carriers of the antigen. By 1978, data were sufficient to permit testing in a clinical trial.

The first subject was inoculated in November 1978, and by October 1979, recruitment had ended. In May 1980, all trial events were reviewed and classified by an expert panel. In June 1980 the code of vaccine and placebo allocation was broken.

DESIGN NARRATIVE:

Randomized, double blind, fixed-sample. A total of 549 subjects were allocated to the vaccine group in which they were treated with highly purified formalin-inactivated virus subunits derived from the plasma of chronic carriers of hepatitis B. A total of 534 were allocated to the placebo group. Both groups received injections at 0, 1 month, and 6 months unless evidence of infection developed before the series was completed.

ELIGIBILITY:
Men at high risk for hepatitis B virus infection, 36 years of age or younger, no recent symptoms of hepatitis, blood specimen negative for HBsAg, anti-HBs and anti-HBe.

Ages: 18 Years to 36 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1978-11; Study Completion 1980-06 (Actual)

REFERENCES:
- [Background] Szmuness W, Stevens CE, Harley EJ, Zang EA, Oleszko WR, William DC, Sadovsky R, Morrison JM, Kellner A. Hepatitis B vaccine: demonstration of efficacy in a controlled clinical trial in a high-risk population in the United States. N Engl J Med. 1980 Oct 9;303(15):833-41. doi: 10.1056/NEJM198010093031501. PMID 6997738